CLINICAL TRIAL: NCT01059773
Title: An Exploratory Trial to Assess Naturalistic Safety and Efficacy Outcomes in Patients With Moderate to Severe Plaque Psoriasis Transitiioned to Ustekinumab From Previous Methotrexate Therapy (TRANSIT)
Brief Title: A Safety and Efficacy Study of Ustekinumab in Patients With Plaque Psoriasis Who Have Had an Inadequate Response to Methotrexate
Acronym: TRANSIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR016639; CR016639 (Registry Identifier: ClinicalTrials.gov); CNTO1275PSO4004 (Other: Janssen CTMS ID)
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Results first posted 2012-01-30 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Psoriasis
Keywords: Psoriasis; Ustekinumab; Stelara; Methotrexate; Biologic
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Methotrexate Cessation (Experimental): Patients will receive ustekinumab by SC injection at Weeks 0, 4, 16, 28 and 40. The last dose of methotrexate will be taken anytime in the week prior to baseline (week 0).
  Interventions: Drug: Ustekinumab
- Gradual Reduction of Methotrexate (Active Comparator): Patients will receive ustekinumab by SC injection at Weeks 0, 4, 16, 28 and 40. Patients will gradually reduce the dose of methotrexate over the 4 week period after week 0.
  Interventions: Drug: Ustekinumab; Drug: Methotrexate

INTERVENTIONS:
Drug: Ustekinumab — Patients weighting ≤ 100 kg will receive ustekinumab 45 mg at Weeks 0, 4 and 16. Patients who achieve a PASI 75 response at Week 28 and 40 will continue receiving ustekinumab 45 mg at Week 28 and 40. Patients who fail to achieve PASI 75 response at Week 28 will receive ustekinumab 90 mg at Week 28 and 40. Patients who achieve a PASI 75 response at Week 28, but fail to achieve PASI 75 response at Week 40 will receive ustekinumab 90 mg at Week 40. Patients > 100 kg will receive ustekinumab 90 mg at Weeks 0, 4, 16, 28 and 40, regardless of achievement of PASI 75 response. Consideration will be given to discontinuing treatment in these patients if they show no response at Week 28.
Drug: Methotrexate — Gradual reduction of methotrexate therapy over the 4 week period after Week 0. The methotrexate dose reduction regime will depend on the dose of methotrexate at screening. All patients will stop methotrexate regardless of the final dose after 4 overlapping weeks. The last dose of methotrexate will be given within the 7 day period before the second dose of ustekinumab.
  Arms: Gradual Reduction of Methotrexate

SUMMARY:
This purpose of this study is to assess the safety of ustekinumab in psoriasis patients who receive ustekinumab following an inadequate response to methotrexate therapy. The study will provide information for doctors on how to manage the transfer from methotrexate to the biologic agent ustekinumab. The study is designed to compare two methods of transferring patients from methotrexate to ustekinumab. The two methods being compared are discontinuation of methotrexate with immediate initiation of ustekinumab versus initiation of ustekinumab with overlap and gradual dose reduction of methotrexate over 4 weeks.

DETAILED DESCRIPTION:
Only limited data exist to guide physicians on transitioning patients onto biologic agents once conventional systemic agents have been found to be inadequate. Most Phase III regulatory studies for biologics, including ustekinumab, required washout periods of between one and three months between previous therapies and the start of study agent. Although advantageous from a methodological perspective, this approach does not appear to mirror real-world clinical practice, in which clinicians and patients are unwilling to go without treatment for extended periods. As a result, physicians appear to employ several arbitrary strategies when transitioning their patients. Two commonly used approaches are: Initiation of biologic therapy with immediate cessation of previous conventional systemic therapy or Initiation of biologic therapy with overlap and gradual reduction of previous conventional systemic therapy. Some physicians opt for the first strategy to minimise the risk of drug-drug interactions. Others opt for the second strategy to minimise the risk of symptomatic worsening between cessation of previous treatment and the onset of action of biologic agents. This study aims to compare safety, efficacy and quality of life outcomes associated with these two strategies, with follow-up for 52 weeks. The primary objective of this exploratory trial is to evaluate the comparative safety through week 12 of two treatment transition strategies in patients with inadequate response to methotrexate: discontinuation of methotrexate with immediate initiation of ustekinumab versus initiation of ustekinumab with overlap and gradual dose reduction of methotrexate over 4 weeks. Secondary objectives of the study include evaluating the safety, efficacy, and quality of life through Week 52. The focus of the trial is on estimation rather than on hypothesis testing and, therefore, no formal hypothesis testing is planned. The primary endpoint is the proportion of patients experiencing one or more treatment-emergent adverse events (AEs) through Week 12 within each treatment transition arm. All proportions will be accompanied by an estimated 95% confidence interval. This is a phase IIIB/IV multicentre, open label, two-arm, randomised study, lasting 56 weeks (including a screening period). The primary endpoint is assessed after 12 weeks of treatment (Week 12). All treated patients will be followed for safety and efficacy through Week 52. Patients will be stratified according to their body weight to ensure a similar distribution of patients >100 kg between the two treatment arms. Approximately 4 weeks prior to study start, all patients who provide consent for participation will be screened according to the requirements of the inclusion and exclusion criteria. Patients who meet all of the inclusion criteria and none of the exclusion criteria will enter the study. During the Screening Phase, patients will continue their current treatment schedule and dose for methotrexate, with folic acid if prescribed. At Week 0, prior to the first dose of ustekinumab, patients will be randomised 1:1 to one of the two treatment arms described below. Patients will be stratified according to their baseline body weight (=<100 kg or >100 kg) to ensure a similar distribution of patients >100 kg between the two treatment arms. Patients eligible for the study will be men and women aged 18 years or older with moderate to severe plaque psoriasis who have a Psoriasis Area and Severity Index (PASI) >=10, who have failed or are intolerant to methotrexate therapy. Patients entering the study must be receiving methotrexate at a dose of 10-25 mg/week, and should have been receiving methotrexate for at least 8 weeks prior to screening. Approximately 576 patients will be included in the study from approximately 100 sites in 20 countries. In both treatment arms, Patients weighing ≤ 100 kg will receive ustekinumab 45 mg at Weeks 0, 4 and 16. Patients who achieve a PASI 75 response at Week 28 and 40 will continue receiving ustekinumab 45 mg at Week 28 and 40. Patients who fail to achieve PASI 75 response at Week 28 will receive ustekinumab 90 mg at Week 28 and 40. Patients who achieve a PASI 75 response at Week 28, but fail to achieve PASI 75 response at Week 40 will receive ustekinumab 90 mg at Week 40. Patients > 100 kg will receive ustekinumab 90 mg at Weeks 0, 4, 16, 28 and 40, regardless of achievement of PASI 75 response. Consideration will be given to discontinuing treatment in these patients if they show no response at Week 28. At Week 0, all eligible patients will be randomised to one of the following treatment regimens. The methotrexate dose reduction regime will depend on the dose of methotrexate at screening. All patients will stop methotrexate regardless of the final dose after 4 overlapping weeks (Weeks 0, 1, 2 and 3). The last dose of methotrexate will be given within the 7 day period before the second dose of ustekinumab. Safety evaluations will include physical examination, body weight and waist circumference, pregnancy testing, vital signs, clinical laboratory testing with full blood analysis and biochemistry, skin assessment for suspicious malignant lesions, Tuberculosis (TB) assessment, adverse events review and collection. Efficacy evaluations, including Psoriasis Area Severity Index (PASI), Nail Psoriasis Severity Index (NAPSI) and Physician's Global Assessment (PGA), will be carried out. Evaluations to assess changes in quality of life, including the Dermatology Life Quality Index (DLQI), Hospital Anxiety Depression Score (HADS), EuroQol-5 dimensional questionnaire (EQ-5D) and Patient Benefit Index (PBI), will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have diagnosis of plaque-type psoriasis for at least 6 months prior to first administration of study agent (patients with concurrent psoriatic arthritis may be enrolled)
* Moderate-to-severe psoriasis scored as PASI >= 10 at screening and at the time of first administration of ustekinumab
* Should currently receive (and have been receiving for at least 8 weeks directly prior to screening) systemic therapy with methotrexate at a dose of at least 10 mg/week but not exceeding 25 mg/week, with an inadequate response to this treatment (due to either efficacy or tolerability) and, in the judgment of the treating physician and patient, a treatment change is needed
* Women should take adequate birth control measures throughout the study and must agree to continue to use such birth control measures and not to become pregnant or plan to become pregnant for at least 15 weeks after the last dose of ustekinumab and for at least 6 months after the last dose of methotrexate
* Men must be using adequate birth control measures whilst receiving methotrexate and for 6 months after the last dose of methotrexate

Exclusion Criteria:

* Patients should not have non-plaque forms of psoriasis (eg, erythrodermic, guttate, or pustular)
* Should currently (and within 12 months) not receive ciclosporin, fumarates, PUVA, etanercept, efalizumab, infliximab, adalimumab or alefacept or other biologic or systemic therapy (and other therapy as indicated in the protocol)
* Women who are pregnant, breastfeeding, or planning pregnancy (both men and women) while enrolled in the study
* Have previously failed treatment with any therapeutic agent directly targeted at reducing IL-12 or IL-23, including, but not limited to, ustekinumab and ABT-874
* Active or latent Tuberculosis or other chronic or recurrent infectious disease
* Known history of lymphoproliferative disease
* Known malignancy or history of malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (76):
- Vienna, Austria
- Belgium (3):
  - Brussels
  - Ghent
  - Liège
- Bulgaria (2):
  - Pleven
  - Sofia
- Denmark (2):
  - Aarhus
  - Roskilde
- Finland (2):
  - Tampere
  - Turku
- France (15):
  - Chambray-lès-Tours
  - Creil
  - Jarez
  - Lille
  - Marseille
  - Montpellier
  - Nantes
  - Nantes Cedex 01 N/A
  - Nice
  - Paris
  - Pessac
  - Pierre-Bénite
  - Poitiers
  - Rouen
  - Toulouse
- Germany (16):
  - Berlin
  - Dresden
  - Erlangen
  - Essen
  - Frankfurt
  - Göttingen
  - Hamburg
  - Kiel
  - Landau
  - Leipzig
  - Mahlow
  - Marburg
  - München
  - Münster
  - Tÿbingen
  - Witten
- Greece (2):
  - Athens
  - Thessaloniki
- Hungary (2):
  - Debrecen
  - Szeged
- Israel (2):
  - Petah Tikva
  - Tel Aviv
- Lithuania (2):
  - Kaunas
  - Vilnius
- Netherlands (2):
  - Nijmegen
  - Rotterdam
- Norway (2):
  - Oslo
  - Stavanger
- Poland (3):
  - Lodz
  - Poznan
  - Wroclaw
- Portugal (2):
  - Lisbon
  - Porto
- Bratislava, Slovakia
- Spain (6):
  - Alicante
  - Badalona
  - Barcelona
  - Córdoba
  - La Coruÿa N/A
  - Madrid
- Sweden (4):
  - Gothenburg
  - Malmo
  - Solna
  - Uppsala
- United Kingdom (7):
  - Aberdeen
  - Cardiff
  - Craigavon
  - Glasgow
  - London
  - Nottingham
  - Salford

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient received on-study methotrexate only but no ustekinumab and was therefore excluded from the analysis.
Groups:
- UST / MTX Stopped: Patients weighing <=100 kg will receive ustekinumab 45 mg (0.5 ml) by SC injection at Weeks 0, 4 and every 12 weeks until Week 40. Patients weighing >100 kg will receive ustekinumab 90 mg (1 ml) in two SC injections. In Arm 1 patients will have immediate cessation of methotrexate therapy.
- UST / MTX Gradually Withdrawn: Patients weighing <=100 kg will receive ustekinumab 45 mg (0.5 ml) by SC injection at Weeks 0, 4 and every 12 weeks until Week 40. Patients weighing >100 kg will receive ustekinumab 90 mg (1 ml) in two SC injections. In Arm 2 patients will have gradual reduction of methotrexate therapy.
Period: Overall Study
Arm/Group | UST / MTX Stopped | UST / MTX Gradually Withdrawn
Started | 244 | 245
Completed | 224 (Completed is refering to no Discontinuation of Study Agent Through Week 52) | 221 (Completed is refering to no Discontinuation of Study Agent Through Week 52)
Not Completed | 20 | 24
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Pregnancy | 1 | 1
Not completed — Protocol Violation | 6 | 2
Not completed — Physician Decision | 5 | 4
Not completed — Lack of Efficacy | 3 | 3
Not completed — Death | 0 | 1
Not completed — Malignancy including squamous cell skin | 0 | 1
Not completed — Ineligible follow TB screening criteria | 0 | 1
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UST / MTX Stopped | UST / MTX Gradually Withdrawn | Total
Number analyzed (Participants) | 244 | 245 | 489
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (12.1) | 47.3 (12.6) | 46.2 (12.4)
Age, Customized [Number; unit: participants]
  18-29 years | 29 | 20 | 49
  30-39 years | 57 | 48 | 105
  40-49 years | 69 | 75 | 144
  50-59 years | 56 | 60 | 116
  >=60 years | 33 | 42 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 83 | 157
  Male | 170 | 162 | 332
Weight, Categorized [Number; unit: participants]
  <= 100 kg | 195 | 196 | 391
  > 100 kg | 49 | 49 | 98

OUTCOME MEASURES:

1. Secondary Outcome: Rate of Adverse Events (AEs), Serious AEs (SAEs) and Deaths During the Study Period
Description: The number of patients with any of the following Treatment Emergent AEs (TEAEs) were summarized through Week 12 and through Week 52, by treatment arm and body weight category (≤100 kg and >100 kg): AE; SAE and Death.
Time Frame: at week 12, 16, 28 40 and 52
Population: All randomized patients who took at least one dose of study medication and set who had any post-baseline safety information.
Measure: Number; unit: Number of patients
Groups:
- UST / MTX Stopped: Patients <=100 kg: Patients weighing <=100 kg will receive ustekinumab 45 mg (0.5 ml) by SC injection at Weeks 0, 4 and every 12 weeks until Week 40. In Arm 1 patients will have immediate cessation of methotrexate therapy.
- UST / MTX Stopped: Patients >100kg: Patients weighing >100 kg will receive ustekinumab 90 mg (1 ml) in two SC injections. In Arm 1 patients will have immediate cessation of methotrexate therapy.
- UST / MTX Gradually Withdrawn: Patients <=100 kg: Patients weighing <=100 kg will receive ustekinumab 45 mg (0.5 ml) by SC injection at Weeks 0, 4 and every 12 weeks until Week 40. In Arm 2 patients will have gradual reduction of methotrexate therapy.
- UST / MTX Gradually Withdrawn: Patients >100kg: Patients weighing >100 kg will receive ustekinumab 90 mg (1 ml) in two SC injections. In Arm 2 patients will have gradual reduction of methotrexate therapy
Arm/Group | UST / MTX Stopped: Patients <=100 kg | UST / MTX Stopped: Patients >100kg | UST / MTX Gradually Withdrawn: Patients <=100 kg | UST / MTX Gradually Withdrawn: Patients >100kg
Number analyzed (Participants) | 195 | 49 | 196 | 49
Number of patients
  Any TEAE: through week 12 | 116 | 33 | 124 | 34
  Any TEAE: through week 16 | 127 | 35 | 135 | 40
  Any TEAE: through week 28 | 141 | 39 | 147 | 42
  Any TEAE: through week 40 | 149 | 40 | 160 | 44
  Any TEAE: through week 52 | 155 | 40 | 162 | 46
  Any serious TEAE: through week 12 | 5 | 2 | 3 | 3
  Any serious TEAE: through week 16 | 6 | 4 | 6 | 3
  Any serious TEAE: through week 28 | 7 | 4 | 10 | 3
  Any serious TEAE: through week 40 | 10 | 4 | 14 | 3
  Any serious TEAE: through week 52 | 15 | 5 | 15 | 5
  Any Death: through week 12 | 0 | 0 | 0 | 1
  Any Death: through week 16 | 0 | 0 | 0 | 1
  Any Death: through week 28 | 0 | 0 | 0 | 1
  Any Death: through week 40 | 0 | 0 | 0 | 1
  Any Death: through week 52 | 0 | 0 | 0 | 1

2. Secondary Outcome: Rate of Severe AEs, Reasonably Related AEs, and AEs Leading to Discontination During the Study Period
Description: The number of patients with any of the following TEAEs were summarized through Week 12 and through Week 52, by treatment arm and body weight category (≤100 kg and >100 kg): AE with severe intensity; AE or SAE reasonably related to ustekinumab (i.e., AEs classified by the investigator as 'possibly', 'probably', or 'very likely' related to study agent); AE or SAE leading to permanent discontinuation of ustekinumab.
Time Frame: at week 12, 16, 28 40 and 52
Population: as for outcome 1
Measure: Number; unit: Number of patients
Arm/Group | UST / MTX Stopped: Patients <=100 kg | UST / MTX Stopped: Patients >100kg | UST / MTX Gradually Withdrawn: Patients <=100 kg | UST / MTX Gradually Withdrawn: Patients >100kg
Number analyzed (Participants) | 195 | 49 | 196 | 49
Number of patients
  Any severe TEAE: through week 12 | 11 | 2 | 5 | 0
  Any severe TEAE: through week 16 | 11 | 3 | 5 | 0
  Any severe TEAE: through week 28 | 11 | 3 | 7 | 0
  Any TEAE: through week 40 | 14 | 4 | 12 | 1
  Any severe TEAE: through week 52 | 18 | 5 | 13 | 3
  Any TEAE related to UST: through week 12 | 41 | 10 | 43 | 13
  Any TEAE related to UST: through week 16 | 46 | 11 | 46 | 14
  Any TEAE related to UST: through week 28 | 47 | 15 | 49 | 15
  Any TEAE related to UST: through week 40 | 54 | 17 | 60 | 17
  Any TEAE related to UST: through week 52 | 56 | 17 | 60 | 18
  Any Serious TEAE related to UST through week 12 | 0 | 1 | 0 | 0
  Any Serious TEAE related to UST through week 16 | 0 | 1 | 0 | 0
  Any Serious TEAE related to UST through week 28 | 0 | 1 | 1 | 0
  Any Serious TEAE related to UST through week 40 | 0 | 1 | 4 | 0
  Any Serious TEAE related to UST through week 52 | 1 | 1 | 4 | 1
  Permanently discontinued UST due to AE: week 12 | 2 | 1 | 1 | 0
  Permanently discontinued UST due to AE: week 16 | 2 | 2 | 1 | 0
  Permanently discontinued UST due to AE: week 28 | 2 | 2 | 1 | 0
  Permanently discontinued UST due to AE: week 40 | 2 | 2 | 2 | 0
  Permanently discontinued UST due to AE: week 52 | 2 | 2 | 1 | 0

3. Primary Outcome: Number of Patients Experiencing One or More Adverse Events Occurring From Week 0 Through Week 12
Time Frame: from week 0 to week 12
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- UST / MTX Stopped: Patients will receive ustekinumab by SC injection at Weeks 0, 4, 16, 28 and 40. The last dose of methotrexate will be taken anytime in the week prior to baseline (week 0).
- UST / MTX Gradually Withdrawn: Patients will receive ustekinumab by SC injection at Weeks 0, 4, 16, 28 and 40. Patients will gradually reduce the dose of methotrexate over the 4 week period after week 0.
Arm/Group | UST / MTX Stopped | UST / MTX Gradually Withdrawn
Number analyzed (Participants) | 244 | 245
participants | 149 | 158

4. Secondary Outcome: Rate of Infections, Severe Infections and Infections Requiring Oral or Parenteral Antimicrobial Treatment During the Study Period
Description: The number of patients with any of the following TEAEs were summarized through Week 12 and through Week 52, by treatment arm and body weight category (≤100 kg and >100 kg): infections, serious infections, and infections requiring oral or parenteral antimicrobial treatment (infections being considered any event that by the investigator was indicated as infection on the CRF).
Time Frame: at week 12, 16, 28 40 and 52
Population: as for outcome 1
Measure: Number; unit: Number of patients
Arm/Group | UST / MTX Stopped: Patients <=100 kg | UST / MTX Stopped: Patients >100kg | UST / MTX Gradually Withdrawn: Patients <=100 kg | UST / MTX Gradually Withdrawn: Patients >100kg
Number analyzed (Participants) | 195 | 49 | 196 | 49
Number of patients
  Any treatment-emergent (TE) infection: week 12 | 36 | 13 | 42 | 11
  Any TE infection: week 16 | 43 | 14 | 50 | 13
  Any TE infection: week 28 | 55 | 18 | 68 | 19
  Any TE infection: week 40 | 61 | 21 | 76 | 23
  Any TE infection: week 52 | 64 | 22 | 81 | 23
  Any serious TE infection: through week 12 | 0 | 1 | 0 | 0
  Any serious TE infection: through week 16 | 0 | 1 | 0 | 0
  Any serious TE infection: through week 28 | 0 | 1 | 1 | 0
  Any serious TE infection: through week 40 | 0 | 1 | 3 | 0
  Any serious TE infection: through week 52 | 0 | 1 | 3 | 0
  Infection requiring antibiotic treatment: week 12 | 13 | 5 | 12 | 2
  Infection requiring antibiotic treatment: week 16 | 19 | 6 | 15 | 2
  Infection requiring antibiotic treatment: week 28 | 23 | 10 | 22 | 6
  Infection requiring antibiotic treatment: week 40 | 25 | 12 | 31 | 7
  Infection requiring antibiotic treatment: week 52 | 27 | 13 | 32 | 8

5. Secondary Outcome: Rate of Malignancies and Other Events of Clinical Interest (Tuberculosis, Serious Cardiovascular Events, Anaphylactic/Serum Sickness Reaction)
Description: The number of patients with a malignancy and other event of clinical interest (tuberculosis, serious cardiovascular events, anaphylactic/serum sickness reaction) were summarized through Week 12 and through Week 52, by treatment arm and body weight category (≤100 kg and >100 kg)
Time Frame: at week 12, 16, 28 40 and 52
Population: as for outcome 1
Measure: Number; unit: Number of patients
Arm/Group | UST / MTX Stopped: Patients <=100 kg | UST / MTX Stopped: Patients >100kg | UST / MTX Gradually Withdrawn: Patients <=100 kg | UST / MTX Gradually Withdrawn: Patients >100kg
Number analyzed (Participants) | 195 | 49 | 196 | 49
Number of patients
  Any treatment-emergent (TE) malignancy: week 12 | 0 | 0 | 0 | 0
  Any TE malignancy: week 16 | 0 | 0 | 0 | 0
  Any TE malignancy: week 28 | 0 | 0 | 2 | 0
  Any TE malignancy: week 40 | 0 | 0 | 2 | 0
  Any TE malignancy: week 52 | 2 | 0 | 2 | 0
  Any TE tuberculosis: through week 12 | 0 | 0 | 0 | 0
  Any TE tuberculosis: through week 16 | 0 | 0 | 0 | 0
  Any TE tuberculosis: through week 28 | 0 | 0 | 0 | 0
  Any TE tuberculosis: through week 40 | 0 | 0 | 0 | 0
  Any TE tuberculosis: through week 52 | 0 | 0 | 0 | 0
  Any TE serious cardiovascular event: week 12 | 0 | 0 | 0 | 0
  Any TE serious cardiovascular event: week 16 | 0 | 0 | 0 | 0
  Any TE serious cardiovascular event: week 28 | 0 | 0 | 0 | 0
  Any TE serious cardiovascular event: week 40 | 0 | 0 | 1 | 0
  Any TE serious cardiovascular event: week 52 | 0 | 0 | 1 | 1
  TE anaphylactic/serum sickness reaction: week 12 | 0 | 0 | 0 | 0
  TE anaphylactic/serum sickness reaction: week 16 | 0 | 0 | 0 | 0
  TE anaphylactic/serum sickness reaction: week 28 | 0 | 0 | 0 | 0
  TE anaphylactic/serum sickness reaction: week 40 | 0 | 0 | 0 | 0
  TE anaphylactic/serum sickness reaction: week 52 | 0 | 0 | 0 | 0

6. Secondary Outcome: Change in Mean Psoriasis Area-and-severity Index (PASI) Score Compared to Baseline
Description: Change from baseline in Psoriasis Area and Severity Index (PASI) (0 [best] - 72 [worst]). The PASI is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score.
Time Frame: at Weeks 0, 2, 4, 12, 16, 28, 40 and 52
Population: The modified intent-to-treat (mITT) analysis includes all subjects who were randomized and received at least one dose of ustekinumab, regardless of their compliance with the protocol. Subjects who dropped out after randomization and before the first administration of ustekinumab were excluded from the mITT analysis
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- UST / MTX Gradually Withdrawn: Patients <=100 kg: Patients will receive ustekinumab by SC injection at Weeks 0, 4, 16, 28 and 40. Patients will gradually reduce the dose of methotrexate over the 4 week period after week 0.
Arm/Group | UST / MTX Stopped | UST / MTX Gradually Withdrawn: Patients <=100 kg
Number analyzed (Participants) | 244 | 243
Units on a scale
  week 2 | -3.73 (4.69) | -4.28 (4.37)
  week 4 | -7.65 (5.93) | -7.82 (5.42)
  week 12 | -12.93 (7.35) | -12.7 (6.6)
  week 16 | -12.84 (7.44) | -12.97 (7.11)
  week 28 | -13.38 (7.8) | -13.43 (7.47)
  week 40 | -13.78 (7.65) | -13.47 (6.61)
  week 52 | -13.84 (7.24) | -13.98 (6.62)

7. Secondary Outcome: Proportion of Patients Achieving PASI 50 Response
Description: This is based on the number of participants achieving at least 50% improvement from baseline in Psoriasis Area and Severity Index (PASI) (0 [best] - 72 [worst]). The PASI is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score.
Time Frame: at Weeks 2, 4, 12, 16, 28, 40 and 52
Population: The modified intent-to-treat (mITT) analysis set includes all subjects who were randomized and received at least one dose of ustekinumab, regardless of their compliance with the protocol. Subjects who dropped out after randomization and before the first administration of ustekinumab were excluded from the mITT analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | UST / MTX Stopped | UST / MTX Gradually Withdrawn
Number analyzed (Participants) | 244 | 243
Percentage of participants
  week 2 | 10.3 [6.5 to 14.1] | 15.6 [11.1 to 20.2]
  week 4 | 39.3 [33.1 to 45.4] | 49.2 [42.9 to 55.5]
  week 12 | 83.8 [79.2 to 88.5] | 86.1 [81.7 to 90.5]
  week 16 | 83.5 [78.7 to 88.2] | 84.2 [79.5 to 88.8]
  week 28 | 84.9 [80.3 to 89.5] | 87.7 [83.5 to 91.9]
  week 40 | 90.7 [86.9 to 94.5] | 88.5 [84.3 to 92.7]
  week 52 | 90.6 [86.8 to 94.4] | 91.0 [87.2 to 94.7]

8. Secondary Outcome: Proportion of Patients Achieving PASI 75 Response
Description: This is based on the number of participants achieving at least 75% improvement from baseline in Psoriasis Area and Severity Index (PASI) (0 [best] - 72 [worst]). The PASI is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score.
Time Frame: at Weeks 2, 4, 12, 16, 28, 40 and 52
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | UST / MTX Stopped | UST / MTX Gradually Withdrawn
Number analyzed (Participants) | 244 | 243
Percentage of participants
  week 2 | 2.9 [0.8 to 5.0] | 2.5 [0.5 to 4.4]
  week 4 | 12.0 [7.9 to 16.1] | 15.3 [10.8 to 19.8]
  week 12 | 58.1 [51.9 to 64.3] | 62.2 [56.0 to 68.3]
  week 16 | 63.6 [57.4 to 69.7] | 64.6 [58.5 to 70.6]
  week 28 | 71.1 [65.3 to 77.0] | 71.1 [65.3 to 76.9]
  week 40 | 76.9 [71.4 to 82.4] | 72.1 [66.3 to 78.0]
  week 52 | 76.3 [70.8 to 81.9] | 76.9 [71.4 to 82.5]

9. Secondary Outcome: Proportion of Patients Achieving PASI 90 Response
Description: This is based on the number of participants achieving at least 90% improvement from baseline in Psoriasis Area and Severity Index (PASI) (0 [best] - 72 [worst]). The PASI is a test of how bad a person's psoriasis is. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score.
Time Frame: at Weeks 2, 4, 12, 16, 28, 40 and 52
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | UST / MTX Stopped | UST / MTX Gradually Withdrawn
Number analyzed (Participants) | 244 | 243
Percentage of participants
  week 2 | 0.4 [0.0 to 1.2] | 0.8 [0.0 to 2.0]
  week 4 | 3.3 [1.1 to 5.6] | 3.3 [1.1 to 5.6]
  week 12 | 33.2 [27.2 to 39.1] | 31.9 [26.0 to 37.9]
  week 16 | 39.0 [32.8 to 45.2] | 42.1 [35.8 to 48.3]
  week 28 | 46.6 [40.1 to 53.0] | 47.7 [41.3 to 54.0]
  week 40 | 46.7 [40.1 to 53.2] | 49.1 [42.6 to 55.6]
  week 52 | 47.8 [41.2 to 54.3] | 49.3 [42.7 to 55.9]

ADVERSE EVENTS:
Time Frame: From week 0 to week 52
Description: Only subjects who had at least one of the TEAEs listed in the Other (non Serious) AE table are included in the Total no. subjects with Non-Serious Adverse Events.
Arm/Group | UST / MTX Stopped | UST / MTX Gradually Withdrawn
Serious Adverse Events (participants affected / at risk) | 20/244 | 20/245
Other Adverse Events (participants affected / at risk) | 113/244 | 132/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UST / MTX Stopped (N=244) | UST / MTX Gradually Withdrawn (N=245)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 2 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Alcoholism (Psychiatric disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Femoral artery occlusion (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UST / MTX Stopped (N=244) | UST / MTX Gradually Withdrawn (N=245)
Nasopharyngitis (Infections and infestations) | 49 | 57
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 14
Headache (Nervous system disorders) | 33 | 33
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 17
Psoriasis (Skin and subcutaneous tissue disorders) | 9 | 20
Hypertension (Vascular disorders) | 16 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the Sponsor for review at least 60 days prior to submission for publication or presentation. No paper that incorporates Confidential Information will be submitted for publication without Sponsor's prior written consent. If requested in writing, such publication will be withheld for up to an additional 60 calendar days. A publication from the individual Study site data will not be published until the combined results have been published.